CLINICAL TRIAL: NCT01918111
Title: Effects of REnal Denervation for Resistant Hypertension on Exercise Diastolic Function and Regression of Atherosclerosis and the Evaluation of NEW Methods Predicting A successfuL Renal Sympathetic Denervation (RENEWAL-EXERCISE, -REGRESS, and -PREDICT Trial From RENEWAL RDN Registry)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study terminated early due to the difficulty of recruiting candidates.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0025
Record Dates: First submitted 2013-07-09; First posted 2013-08-07 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2016-12

CONDITIONS: Resistant Hypertension
Keywords: Renal denervation, Exercise diastolic function, Atherosclerosis, New methods
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RD group (Experimental): Renal denervation group
  Interventions: Procedure: Renal denervation
- Control group (Active Comparator): Control group
  Interventions: Drug: adenosine infusion treatment

INTERVENTIONS:
Procedure: Renal denervation — Renal denervation will be performed via common femoral artery with standard endovascular technique and simplicity catheter
  Arms: RD group
Drug: adenosine infusion treatment — Continue hypertensive medication
  Arms: Control group

SUMMARY:
1. (RENEWAL-EXERCISE trial) The investigators hypothesize that the increased sympathetic nervous system activation that is associated with resistant hypertension is a major contributor in the pathogenesis of exercise diastolic dysfunction and that modulation of the sympathetic nervous system activity with radiofrequency ablation of the renal artery sympathetic nerve fibers delivered via a treatment catheter, will have a significant effect on the diastolic function that is beyond BP-lowering effect.
2. (RENEWAL-REGRESSION trial) The major cause of mortality and morbidity in hypertension is atherosclerotic cardiovascular disease. the significant decrease in the sympathetic nervous system activation after renal sympathetic denervation will contribute to regression over and beyond it's effect of blood pressure reduction.
3. (RENEWAL-PREDICT trial) No data exists regarding the tests or methods predicting the successful renal denervation causing the effective reduction of BP. For these, the investigators sought to perform the new tests such as adenosine infusion test during procedure and skin sympathetic activity measurement before and immediate post-procedure (detailed explanation provided in section of Methods) and then evaluate the association between these tests and reduction of BP following procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-85 years with resistant hypertension defined as systolic BP>140 mmHg (>130 mmHg for diabetes) or diastolic BP>90mmHg (>80 mmHg for diabetes) despite adequate administration of 3 or more different classes of anti-hypertensive medications including diuretics with good adherence and adequate treatment regimen.
* All agents should be prescribed at optimal dose amounts. BP was based on an average of 3 office BP readings measured according to the general guidelines. Patients are adhering to a stable drug regimen including 3 or more antihypertensive medications (with no changes for a minimum of 2 weeks prior to enrollment).
* Patients provided with the written, informed consent to participate in this study

Exclusion Criteria:

* Hemodynamically or anatomically significant renal artery abnormalities, main renal arteries < 4 mm in diameter or < 20 mm in length, or.prior renal artery intervention
* Estimated glomerular filtration rate (eGFR) of < 30mL/min/1.73m2, using the MDRD calculation
* Hemodynamically significant valvular heart disease
* History of congestive heart failure with reduce LV ejection fraction of less than 35%
* CVA in the prior 3 months
* ST-segment elevation MI within 48 hours
* Scheduled or planned surgery or cardiovascular intervention in the next 6 months.
* Patients with chronic debilitating disease with life expectancy of less than 1 year
* Patients taking hormone replace treatment and/or oral contraceptives; pregnant, nursing or planning to be pregnant
* Chronic liver cirrhosis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
Change in coronary atheroma | change in coronary atheroma for 24 months after renal denervation
  Evaluation of the change in coronary atheroma (change in percent atheroma volume (PAV) and the change in nominal atheroma volume in the 10-mm subsegment with the greatest disease severity at baseline), analyzed by an IVUS, between baseline and 2-year IVUS in the patients with CAD) for RENEWAL-REGRESS trial

SECONDARY OUTCOMES:
Reduction of peak exercise E/E prime | Peak exercise E/E prime from 6 and 12 months after renal denervation
  Reduction of peak exercise E/E prime at 6 month follow up for RENEWAL-EXERCISE trial

OTHER OUTCOMES:
Evaluation of the novel methods predicting the successful renal sympathetic denervation after RDN | change of blood pressure at 6 and 12 months
  Evaluation of the novel methods predicting the successful or unsuccessful renal sympathetic denervation after RDN: 1) Effects the change of blood pressure by infusion of intra-renal adenosine at pre- and immediate post-RND on blood pressure at 6 and 12 months; 2) Association of skin sympathetic activity measurement before and immediate post-procedure and blood pressure at 6 and 12 months; RENEWAL-PREDICT trial)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Pisano A, Iannone LF, Leo A, Russo E, Coppolino G, Bolignano D. Renal denervation for resistant hypertension. Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD011499. doi: 10.1002/14651858.CD011499.pub3. PMID 34806762